CLINICAL TRIAL: NCT06032793
Title: Effects of Deep Breathing Exercise on Pulmonary Function, Perceived Stress and Physical Fitness Among Healthy Smokers.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/MS-PT/01656 Talliya Naz
Record Dates: First submitted 2023-09-05; First posted 2023-09-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Cigarette Smoking
MeSH Terms: conditions — Cigarette Smoking | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep breathing exercise (Experimental): This group will perform following exercises:
  Pursed lip breathing, Diaphragmatic breathing and powered breathing for 3-4 times a day for 6 weeks.
  Interventions: Other: Breathing exercises
- No Intervention (No Intervention): This group will not perform any exercise.

INTERVENTIONS:
Other: Breathing exercises — Pursed lip breathing, Diaphragmatic breathing and powered breathing
  Arms: Deep breathing exercise

SUMMARY:
Effects of deep breathing exercise on pulmonary function, perceived stress and physical fitness among healthy smokers.

DETAILED DESCRIPTION:
Smoking is injurious to health as cigarette contains harmful substances that cause different life threatening diseases, like bronchitis, asthma, chronic obstructive pulmonary disease (COPD), cardiovascular diseases etc. During normal breathing, oxygen is supplied to the body through blood circulation. But, in smokers, carbon monoxide (CO) is supplied to body instead of oxygen, resulting in respiratory issues, like breathlessness and coughing, in acute stages . Smoking decreases lung capacity, as it contains acidic substances which start damaging the lining of the bronchi and bronchioles due to which they become inflamed and infected, resulting into coughing, shortness of breath and chest pain that leads towards chronic bronchitis. This study will contribute our young smokers as they are adherent to smoking and its difficult for them to quit smoking. as their physical activity is limited, individuals under stress condition and with pulmonary complications so impact of this research is that along with helping smokers to quit smoking also applying alternative strategies to minimize complication and improve quality of life. and these alternative strategies include such activities that performed easily at home and do not require much effort or no need to go to gym or any other place to perform these exercises.

ELIGIBILITY:
Inclusion Criteria:

* Only Male Healthy Smoker.
* Age: 20 - 30 years.
* Participants had a minimum smoking history of 5 years.
* Subject without any chronic pulmonary complication.

Exclusion Criteria:

* Smokers with any pulmonary disease, acute infections, other systemic disease.
* Chest deformity or any disability.
* History of any surgery.
* Not willing to participate.

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only male participants
Enrollment: 52 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Forced Vital Capacity | baseline, on 2nd ,4th and 6th week
  The volume of air which can be forcefully expelled from the lungs after taking a deep breath is known as forced vital capacity (FVC). The normal range of FVC for an adult lies between 3.0 and 5.0 L (29). The participant will be asked to seal their lips tightly over the mouthpiece and inhale as deeply as possible. Then they will exhale as forcefully as they can.
Forced Expiratory Volume | baseline, on 2nd ,4th and 6th week
  FEV1 assesses how much air an individual can forcefully exhale. The forced expiratory volume in 1 second (FEV1) is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration. The forced expiratory volume (FEV) can be calculated for the first, second, and/or third seconds of the forced breath. With reference to GOLD range of COPD, the normal value for FEV is <80. An FEV1 of less than 1 L indicates significant lung disease. For correct measures, the procedure will be repeated 3 times, and then the best value will be taken. The FEV1 is the measurement of dynamic volume most often used in conjunction with the FVC in analysis of spirometry.
PERCEIVED STRESS | baseline, on 2nd ,4th and 6th week
  A more precise measure of personal stress can be determined by using a variety of instruments that have been designed to help measure individual stress levels. The first of these is called the Perceived Stress Scale. The Perceived Stress Scale (PSS) is a classic stress assessment instrument. It was originally developed in 1983.
Physical Fitness | baseline, 2nd, 4th and on 6th week
  The six minute walking test (6MWT) will be used to determine the physical fitness. Each patient will be administered a 6-minute walk test. Two cones will be placed 100 feet apart in a hallway. Patients will instructed to walk as many laps around the cones as possible. A calibrated electronic pedometer (Omron Health Care Corporation, Vernon Hills, IL) will be worn on the hip of each patient to obtain the total number of steps taken during the test. Researcher will stand at the center of the 100-foot course and will encourage the patient after every 2 minutes. The researcher will record the time and distance to onset of exhaustion as well as the total distance walked and the total number of steps taken during the test. The walking distances will be subsequently converted from feet to meters.

SECONDARY OUTCOMES:
Sleep quality | baseline, 2nd, 4th and on 6th week
  To determine the sleep quality, Pittsburgh Sleep Quality Index (PSQI) will be used. It was designed to evaluate overall sleep quality in the populations with an internal reliability of a = .83, a test-retest reliability of .85 for the global scale, a sensitivity of 89.6%, and a specificity of 86.5%. Each of the questionnaire's 19 self-reported items belongs to one of seven subcategories: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction.

CONTACTS AND LOCATIONS:
Overall Officials: Malik Muhammad Ali Awan, MSPT, Principal Investigator — Riphah International University, Islamabad
Locations (1):
- Railway General Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No